CLINICAL TRIAL: NCT05775588
Title: Long-term Effects of Endobronchial Valve Implantation on Cardiac Function and Skeletal Muscle Function in Patients With Lung Volume Reduction Surgery
Brief Title: Long-term Effects of Endobronchial Valve Implantation on Cardiac Function and Skeletal Muscle Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-NHLHCRF-LX-01-0202-1
Record Dates: First submitted 2023-02-23; First posted 2023-03-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung volume reduction surgery group (Experimental)
  Interventions: Procedure: Lung volume reduction surgery with endobronchial valve implantation

INTERVENTIONS:
Procedure: Lung volume reduction surgery with endobronchial valve implantation — the patient would undergo Lung volume reduction surgery with endobronchial valve implantation

SUMMARY:
The goal of this type of study: clinical trial is to evaluate the effect of bronchial valve implantation on cardiac function and skeletal muscle function in Chronic Obstructive Pulmonary Disease. The main question it aims to answer are:evaluate the effect of bronchial valve implantation on cardiac function and skeletal muscle function.

Participants will undergo Lung volume reduction surgery with endobronchial valve implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Obstructive Pulmonary Disease
* FEV1 ≤ 45% pred and FEV1/FVC<70%
* TLC>100% pred and RV>175% pred
* CAT score≥18
* Emphysema damage>50%
* Complete interlobar fissure >95% based on quantitative analysis of CT measurement
* No smoking>6 months
* Sign the informed consent form

Exclusion Criteria:

* PaCO2>8.0 kPa, or PaO2<6.0 kPa
* 6-minute walk test<160m
* Obvious chronic bronchitis, bronchiectasis or other infectious pulmonary diseases
* More than 3 hospitalizations for pulmonary infection in the past 12 months before baseline assessment
* Previous lobectomy, LVRS or lung transplantation
* LVEF<45% and or RVSP>50mmHg
* Anticoagulant therapy that cannot be stopped before surgery
* Patients with obvious immune deficiency
* Participated in other lung drug studies within the first 30 days of this study
* Pulmonary nodules requiring intervention
* Any disease or condition that interferes with the completion of the initial or subsequent assessment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline ventricular volume | Baseline
  cardiac magnetic resonance imaging
Ventricular volume （6 months after surgery） | 6 months after surgery
  cardiac magnetic resonance imaging
Ventricular volume（12 months after surgery） | 12 months after surgery
  cardiac magnetic resonance imaging
Baseline FEV1 | Baseline
  Pulmonary function tests
FEV1 （6 months after surgery） | 6 months after surgery
  Pulmonary function tests
FEV1（12 months after surgery） | 12 months after surgery
  Pulmonary function tests
Baseline left Ventricular Ejection Fractions | Baseline
  Echocardiography
Left Ventricular Ejection Fractions （6 months after surgery） | 6 months after surgery
  Echocardiography
Left Ventricular Ejection Fractions （12 months after surgery） | 12 months after surgery
  Echocardiography
Baseline exercise tolerance | Baseline
  6-minute walk test
Exercise tolerance （6 months after surgery） | 6 months after surgery
  6-minute walk test
Exercise tolerance （12 months after surgery） | 12 months after surgery
  6-minute walk test
Baseline health impairment and quality of life of patients Baseline health impairment and quality of life of patients | Baseline
  St. George's Respiratory Questionnaire
Health impairment and quality of life of patients （6 months after surgery） | 6 months after surgery
  St. George's Respiratory Questionnaire
Health impairment and quality of life of patients （12 months after surgery） | 12 months after surgery
  St. George's Respiratory Questionnaire
Baseline cross sectional area of rectus femoris | Baseline
  Rectus femoris ultrasound
Cross sectional area of rectus femoris （6 months after surgery） | 6 months after surgery
  Rectus femoris ultrasound
Cross sectional area of rectus femoris （12 months after surgery） | 12 months after surgery
  Rectus femoris ultrasound
Baseline mmuscle strength of lower limb | Baseline
  Myometer
Mmuscle strength of lower limb （6 months after surgery） | 6 months after surgery
  Myometer
Mmuscle strength of lower limb （12 months after surgery） | 12 months after surgery
  Myometer

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China